CLINICAL TRIAL: NCT05044312
Title: Sleep Disturbances in Surgical Patients With GI Cancers: A Quantitative and Qualitative Analysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI requested
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2019-1182; NCI-2021-09807 (Other: Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2021-09-09; First posted 2021-09-14 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: GI Cancers; Gastrointestinal Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Disturbances (Other): Difficulty Sleeping
  Interventions: Other: Sleeping Disturbances

INTERVENTIONS:
Other: Sleeping Disturbances — most common complaints of patients after surgery and may affect the ability to carry out daily activities, quality of life, and post-surgery recovery.

SUMMARY:
The primary objective of the study is to determine sleep disturbance and its types among patients with gastrointestinal cancers during the perioperative period (preoperative and in-hospital stay following surgery) by using Richard Campbell sleep questionnaire (RCSQ).

The primary objective of this study is to determine the SD during preoperative and post-operative periods evaluated by Richard Campbell Sleep questionnaire. Patients will be asked every 24 hours while at the hospital (before and after surgery) to fill out this questionnaire. The mean RCSQ score at each time point (i.e., before and after surgery) will be calculated for each patient. The overall mean (across all patients) will be calculated and reported along a 95% CI.

DETAILED DESCRIPTION:
Primary:

• Determine sleep disturbance and its types among patients with gastrointestinal cancers during the perioperative period (preoperative and in-hospital stay following surgery) by using Richard Campbell sleep questionnaire(RCSQ).

Secondary:

* Determine sleep disturbance and its types at 30 day post-discharge follow-up visit by RCSQ.
* Determine the correlation between objective sleep variables assessed using Actigraphy and Fitbit and patient-reported SD on Richard Campbell Sleep questionnaire.
* Determine the association of severity and impact of SD among Quality of recovery (QoR-15), Pittsburgh sleep quality index, MDASI-GI and Richard Campbell Sleep questionnaire, and Insomnia Severity Index (ISI).

Exploratory:

• Determine the association between the preoperative inflammatory burden, sleep health {insomnia (using Insomnia Severity Index (ISI)),sleep architecture(sleep-wake cycles usingActigraphy)}, and perioperative inflammatory responses on postoperative SD

ELIGIBILITY:
Inclusion Criteria:

1. Adult GI Cancer patients admitted for elective gastrointestinal surgery.
2. Patients with an expected hospitalstay of at least 72 hours.
3. Able to be able to read and speak English.
4. Must have access to internet or use of mobile device for FitBit.

Exclusion Criteria:

1. <18 years of age.
2. Night shift workers. Obtained from job history, any patient >/= 2 days per week, within the last six months prior consenting, are not eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-06 (Estimated); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Correlating the sleep disturbance and its types among patients with gastrointestinal cancers. | through study completion, an average of 1 year
  This questionnaire will be used to assess during the stay by using (preoperative and in-hospital stay following surgery) by using Richard Campbell sleep questionnaire(RCSQ). scale of 1 to 10 (with 1 being "poor" and 10 being "excellent

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Yennu, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT05044312/ICF_000.pdf